CLINICAL TRIAL: NCT04205604
Title: 18F-Fluoro-L- DOPA PET Imaging for the Detection and Localization of Focal Congenital Hyperinsulinism
Brief Title: 18FluoroLDOPA PET Imaging for the Detection and Localization of Focal Congenital Hyperinsulinism
Acronym: DOPA PET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Miguel Pampaloni (Other)
Responsible Party: Sponsor-Investigator, Miguel Pampaloni, Associate Professor of Radiology & Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8F-Fluoro-L- DOPA
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm, (Experimental): Patients with clinically diagnosed congenital hyperinsulinism
  Interventions: Drug: 18F-Fluoro Dopa Imaging

INTERVENTIONS:
Drug: 18F-Fluoro Dopa Imaging — Imaging with 18F-Fluoro Dopa PET Imaging

SUMMARY:
The goal of this project is to determine the role of FDOPA/PET as a pre-operative diagnostic imaging procedure for differentiating focal and diffuse forms of congenital hyperinsulinism and locating focal lesions in the pancreas to guide surgical resection.

DETAILED DESCRIPTION:
Congenital hyperinsulinism (HI) is the most common cause of recurrent and persistent hypoglycemia, presenting early in infancy. Patients who fail medical therapy usually require resection of the diseased pancreas(partial or subtotal pancreatectomy) to control this disorder. Over half of patients undergoing surgery have a focal area of islet cell dysfunction that is curable with resection. These focal lesions are areas of adenomatosis consisting of a clone of beta-cells that express a paternally-derived mutation of the KATP channel due to loss of heterozygosity for the maternal allele. Current imaging techniques cannot differentiate focal and diffuse forms of hyperinsulinism, nor can they locate focal areas of disease within the pancreas before surgery. L-DOPA is taken up by some neuroendocrine cells, including pancreatic islet cells, and stored as dopamine in secretory granules. Recent studies show that positron emission tomography (PET) following administration of 18F-fluoro-L-DOPA (FDOPA) can distinguish focal and diffuse forms of HI and accurately locate focal lesions within the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Any age, but primarily infants 0-6 months given typical age of initial presentation.
* Children with diagnosis of FoHI or DiHI based on clinical criteria (fasting hypoglycemia accompanied by inadequate suppression of plasma insulin, inappropriately low plasma free fatty acid and plasma-hydroxybutyrate concentrations, and an inappropriate glycemic response to glucagon injection)

  o confirmed by genetic testing for mutations in ABCC8 and KCNJ1 was1.
* Hypoglycemia uncontrolled with medical management (diazoxide, octreotide).
* Able to withdraw medications in time to wash out prior to the scheduled PET scan.
* Patients fulfilling criteria above but with uncontrolled hypoglycemia after initial surgical management (partial or near-total pancreatectomy)
* Normal hepatic and renal function.

Exclusion Criteria:

* Treatment with other, third-line, medications for hyperinsulinism (nifedipine, glucagon).
* Patients with hepatic or renal insufficiency.

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Imaging | four weeks
  To determine the sensitivity and specificity of FDOPA PET/CT in differentiating focal and diffuse forms of HI in infants with medically refractory hypoglycemia
Accuracy of Imaging | four weeks
  To determine the accuracy of FDOPA PET/CT localizing areas of islet cell adenomatosis within the pancreas in patients with focal HI, by identifying the area of abnormal uptake of the raioligand

SECONDARY OUTCOMES:
Semiquantitative Imaging Assessment | four weeks
  o determine whether data from FDOPA PET/CT can accurately quantify pancreatic islet cell mass in patients with HI (normal pancreas, areas of adenomatosis in focal HI and diseased pancreas in diffuse HI) by quantifying the standardized uptake value (SUV) of FDOPA of and correlating with histologic findings.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Hernandez Pampaloni, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No